CLINICAL TRIAL: NCT03127800
Title: The Effect of Acute Intravenous Morphine Administration on Sleep Disordered Breathing (SDB) in Patients With Moderate Obstructive Sleep Apnoea (OSA): A Paired Design Trial
Brief Title: Morphine in Moderate Obstructive Sleep Apnoea
Acronym: MIMOSA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulties with recruitment
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P01911
Record Dates: First submitted 2016-06-13; First posted 2017-04-25 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Obstructive Sleep Apnoea
Keywords: Obstructive Sleep Apnoea; Morphine sulphate; Sleep Disordered Breathing; Central Sleep Apnoea; Hypoxaemia; Hypercapnia; Cheyne-Stokes Respiration; Analgesia; Respiration; Apnoea-Hypopnea Index; Oxygen Desaturation Index; Oximetry; Respiratory Polygraphy; Polysomnography
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep Apnea, Central; Hypoxia; Hypercapnia; Cheyne-Stokes Respiration; Agnosia; Respiratory Aspiration | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Morphine sulphate (Experimental): Participants will be given a first dose of morphine sulphate (intravenously) before bedtime and a second dose four hours later. In both instances 4 mg of intravenous ondansetron will be administered after the morphine sulphate dose to prevent sickness
  Interventions: Drug: Morphine sulphate

INTERVENTIONS:
Drug: Morphine sulphate — 5mg of intravenous morphine sulphate diluted to 5ml with normal saline (0.9% sodium chloride) will be administered 30 minutes before participant's bed time. The same dose will be administered four hours later. In both instances 4 mg of intravenous ondansetron will be administered after the morphine sulphate dose to prevent sickness.
  Other Names: Morphine sulphate 10mg/ml

SUMMARY:
The aim of this study is to investigate the effects of morphine (a drug commonly used for the treatment of moderate to severe pain, particularly following surgery) on the number of pauses in breathing in patients with moderate obstructive sleep apnoea (OSA). Morphine has been shown to reduce upper airway muscle tone and can also cause shallow breathing, which can affect breathing function in patients with sleep apnoea. However, to date these effects have not been proven in clinical trials. Although, caution is advised when prescribing morphine to patients with sleep apnoea, there is currently no strong evidence that morphine makes sleep apnoea worse. Only one randomised controlled trial (considered the gold standard in medical research) has shown no worsening of symptoms for patients with sleep apnoea. The effect of morphine on patients with sleep apnoea will be assessed in a safe, controlled, hospital environment. Information from the study will help inform doctors about the safety of giving morphine to patients with sleep apnoea in urgent situations, for example after surgery.

The results of this study will enable clinicians to make better decisions when prescribing this drug to patients with OSA in the future.

DETAILED DESCRIPTION:
Sleep Disordered Breathing (SDB) is a term used to cover a range of breathing events encountered during sleep and includes Obstructive Sleep Apnoea (OSA). OSA is the most common form of SDB and is caused by partial or complete upper airway occlusion during sleep leading to repetitive arousals to restore the airway patency. These frequent, obstructive events can be associated with symptoms of unrefreshing sleep and adverse health outcomes. The incidence of OSA is increasing due to rising levels of obesity, which has been identified as the strongest risk factor for developing OSA. It is estimated that at present 80% of sufferers are undiagnosed. It must therefore be assumed that some of these patients are referred for surgery.

Morphine, opiates and opioids remain the treatment of choice for moderate and severe pain relief. Inevitably, a large number of patients will be presenting for surgery and receiving postoperative opioid analgesia. Opioids may reduce respiratory rate and tidal volume, decrease chemoresponsiveness to hypercapnia/hypoxia as well as decrease upper airway muscle tone. These effects might further impair respiratory function in patients with SDB. There is limited data showing increased extubation complications, increased incidence of paradoxical breathing patterns and pronounced oxygen desaturations in patients with SDB receiving opioid-based analgesia, but only one randomised controlled trial examining the effect of an opioid in subjects with SDB.

Therefore, the current evidence base regarding the management of patients with OSA and their peri-operative risk is sparse. As such the current recommendation from the American Society of Anaesthesiologists to limit the use of opioids in such patients, is based on expert opinion only. Indeed the effect of opioid analgesia on patients with SDB remains poorly understood, making informed decisions when prescribing such substances to patients with SDB a challenge.

This prospective, paired design trial will investigate the effect of intravenous morphine sulphate on respiration during sleep in patients with moderate OSA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Patients with diagnosis of moderate or severeOSA at screening, diagnosed by nocturnal oximetry, rPSG or PSG (defined as AHI or ODI of 15-50 events/hour) established on Continuous Positive Airway Pressure (CPAP)
3. Patients established on CPAP with confirmed moderate OSA (AHI 15-29 events/hr) 6 nights after withdrawal of CPAP (confirmed at baseline rPSG)
4. Patients diagnosed with moderate OSA by rPSG or PSG, naïve to CPAP treatment

Exclusion Criteria:

* Inability to give informed consent or comply with the protocol
* Current, clinically significant acute respiratory tract infection (at screening and at study visit)
* Chronic respiratory disease (other than OSA), symptomatic ischemic heart disease
* Pregnancy or suspected pregnancy/breast feeding
* Current or recent (within last week of entering the trial and for the duration fo the trial) use of gabapentin, pregabalin, melatonin, mirtazapine, benzodiazepines, barbiturates, sodium oxybate, ramelteon, Z-drugs and opiates/opioids
* Monoamine oxidase inhibitors (MAOIs), linezolid taken within two weeks of participation in the trial
* A known allergy to the investigational medicinal product (IMP) or non investigational medicinal product(s) (NIMP)(s)
* Patients with an inadequate command of English and such that an interpreter would be required overnight
* Change in weight of greater than 5% since the baseline rPSG
* Vital signs recordings (oxygen saturations, blood pressure, pulse rate) that in the clinician's opinion deem the patient unsafe to participate in the trial
* Clinician deems the patient unsafe to participate in the trial (e.g. severely sleepy patients who cannot withdraw from CPAP)
* CPAP intolerant/poor responder
* History of drug abuse (oral and intravenous) including: alcohol, substituted amphetamines, barbiturates, benzodiazepines, cocaine, methaqualone, cannabis and opioids
* A drop of oxygen saturations below 85% continuously for longer than five minutes during the baseline rPSG
* Professional driver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2017-11-04 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Change in Apnoea-Hypopnea Index (AHI) | Change in AHI from baseline Respiratory Polygraphy (rPSG) through to completion of study at overnight visit, within 4 months of baseline
  Change in the mean number of apnoeas and hypopneas.

SECONDARY OUTCOMES:
Change in arterial oxygen desaturations | Change in arterial oxygen desaturations from baseline Respiratory Polygraphy (rPSG) through to completion of study at overnight visit, within 4 months of baseline
  Number of arterial oxygen desaturations of greater than or equal to 4% per hour (Oxygen Desaturation Index) measured by pulse oximetry during the rPSG
Change in the percentage of time spent with nocturnal saturations | Change in percentage of time spent with nocturnal saturations from baseline Respiratory Polygraphy (rPSG) through to completion of study at overnight visit, within 4 months of baseline
  Percentage of time spent with nocturnal saturations of less than or equal to 90% measured by pulse oximetry during the rPSG

CONTACTS AND LOCATIONS:
Overall Officials: Ian Smith, MBBS, Study Director — Papworth Hospital NHS Foundation Trust; Martina Mason, MBBS, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available

REFERENCES:
- [Background] Beloeil H, Delage N, Negre I, Mazoit JX, Benhamou D. The median effective dose of nefopam and morphine administered intravenously for postoperative pain after minor surgery: a prospective randomized double-blinded isobolographic study of their analgesic action. Anesth Analg. 2004 Feb;98(2):395-400. doi: 10.1213/01.ANE.0000093780.67532.95. PMID 14742377
- [Background] Bernards CM, Knowlton SL, Schmidt DF, DePaso WJ, Lee MK, McDonald SB, Bains OS. Respiratory and sleep effects of remifentanil in volunteers with moderate obstructive sleep apnea. Anesthesiology. 2009 Jan;110(1):41-9. doi: 10.1097/ALN.0b013e318190b501. PMID 19104169
- [Background] Boldt J, Thaler E, Lehmann A, Papsdorf M, Isgro F. RETRACTED: Pain management in cardiac surgery patients: comparison between standard therapy and patient-controlled analgesia regimen. J Cardiothorac Vasc Anesth. 1998 Dec;12(6):654-8. doi: 10.1016/s1053-0770(98)90237-3. PMID 9854662
- [Background] Brown KA, Laferriere A, Moss IR. Recurrent hypoxemia in young children with obstructive sleep apnea is associated with reduced opioid requirement for analgesia. Anesthesiology. 2004 Apr;100(4):806-10; discussion 5A. doi: 10.1097/00000542-200404000-00009. PMID 15087614
- [Background] Catley DM, Thornton C, Jordan C, Lehane JR, Royston D, Jones JG. Pronounced, episodic oxygen desaturation in the postoperative period: its association with ventilatory pattern and analgesic regimen. Anesthesiology. 1985 Jul;63(1):20-8. doi: 10.1097/00000542-198507000-00004. PMID 4014768
- [Background] Dimsdale JE, Norman D, DeJardin D, Wallace MS. The effect of opioids on sleep architecture. J Clin Sleep Med. 2007 Feb 15;3(1):33-6. PMID 17557450
- [Background] Duran J, Esnaola S, Rubio R, Iztueta A. Obstructive sleep apnea-hypopnea and related clinical features in a population-based sample of subjects aged 30 to 70 yr. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):685-9. doi: 10.1164/ajrccm.163.3.2005065. PMID 11254524
- [Background] Esclamado RM, Glenn MG, McCulloch TM, Cummings CW. Perioperative complications and risk factors in the surgical treatment of obstructive sleep apnea syndrome. Laryngoscope. 1989 Nov;99(11):1125-9. doi: 10.1288/00005537-198911000-00004. PMID 2530406
- [Background] Gross JB, Bachenberg KL, Benumof JL, Caplan RA, Connis RT, Cote CJ, Nickinovich DG, Prachand V, Ward DS, Weaver EM, Ydens L, Yu S; American Society of Anesthesiologists Task Force on Perioperative Management. Practice guidelines for the perioperative management of patients with obstructive sleep apnea: a report by the American Society of Anesthesiologists Task Force on Perioperative Management of patients with obstructive sleep apnea. Anesthesiology. 2006 May;104(5):1081-93; quiz 1117-8. doi: 10.1097/00000542-200605000-00026. No abstract available. PMID 16645462
- [Background] Kohler M, Stoewhas AC, Ayers L, Senn O, Bloch KE, Russi EW, Stradling JR. Effects of continuous positive airway pressure therapy withdrawal in patients with obstructive sleep apnea: a randomized controlled trial. Am J Respir Crit Care Med. 2011 Nov 15;184(10):1192-9. doi: 10.1164/rccm.201106-0964OC. PMID 21836134
- [Background] Koo, CY. Respiratory effects of opioids in perioperative medicine. The Open Anesthesiology Journal (Suppl 1-M6):23-4. 2011.
- [Background] Kushida CA, Littner MR, Morgenthaler T, Alessi CA, Bailey D, Coleman J Jr, Friedman L, Hirshkowitz M, Kapen S, Kramer M, Lee-Chiong T, Loube DL, Owens J, Pancer JP, Wise M. Practice parameters for the indications for polysomnography and related procedures: an update for 2005. Sleep. 2005 Apr;28(4):499-521. doi: 10.1093/sleep/28.4.499. PMID 16171294
- [Background] Mogri M, Desai H, Webster L, Grant BJ, Mador MJ. Hypoxemia in patients on chronic opiate therapy with and without sleep apnea. Sleep Breath. 2009 Mar;13(1):49-57. doi: 10.1007/s11325-008-0208-4. Epub 2008 Aug 6. PMID 18683000
- [Background] Scottish Intercollegiate Guidelines Network. Management of Obstructive Sleep Apnoea/Hypopnoea Syndrome in Adults. A national clinical guideline. (Guideline Number 73). 2003.
- [Background] Ostermeier AM, Roizen MF, Hautkappe M, Klock PA, Klafta JM. Three sudden postoperative respiratory arrests associated with epidural opioids in patients with sleep apnea. Anesth Analg. 1997 Aug;85(2):452-60. doi: 10.1097/00000539-199708000-00037. No abstract available. PMID 9249130
- [Background] Shaw IR, Lavigne G, Mayer P, Choiniere M. Acute intravenous administration of morphine perturbs sleep architecture in healthy pain-free young adults: a preliminary study. Sleep. 2005 Jun;28(6):677-82. doi: 10.1093/sleep/28.6.677. PMID 16477954
- [Background] American Pain Society. Principles of analgesic use in the treatment of acute pain and cancer pain. 1999.
- [Background] Stradling J, Smith D, Radulovacki M, Carley D. Effect of ondansetron on moderate obstructive sleep apnoea, a single night, placebo-controlled trial. J Sleep Res. 2003 Jun;12(2):169-70. doi: 10.1046/j.1365-2869.2003.00342.x. No abstract available. PMID 12753355
- [Background] Wang D, Teichtahl H, Drummer O, Goodman C, Cherry G, Cunnington D, Kronborg I. Central sleep apnea in stable methadone maintenance treatment patients. Chest. 2005 Sep;128(3):1348-56. doi: 10.1378/chest.128.3.1348. PMID 16162728
- [Background] Webster LR, Choi Y, Desai H, Webster L, Grant BJ. Sleep-disordered breathing and chronic opioid therapy. Pain Med. 2008 May-Jun;9(4):425-32. doi: 10.1111/j.1526-4637.2007.00343.x. PMID 18489633
- [Background] Yarmush J, D'Angelo R, Kirkhart B, O'Leary C, Pitts MC 2nd, Graf G, Sebel P, Watkins WD, Miguel R, Streisand J, Maysick LK, Vujic D. A comparison of remifentanil and morphine sulfate for acute postoperative analgesia after total intravenous anesthesia with remifentanil and propofol. Anesthesiology. 1997 Aug;87(2):235-43. doi: 10.1097/00000542-199708000-00009. PMID 9286886
- [Background] Young T, Evans L, Finn L, Palta M. Estimation of the clinically diagnosed proportion of sleep apnea syndrome in middle-aged men and women. Sleep. 1997 Sep;20(9):705-6. doi: 10.1093/sleep/20.9.705. PMID 9406321
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434